CLINICAL TRIAL: NCT04499105
Title: Effectiveness and Safety of Allogenic Mesenchymal Stem Cell (MSC) Implantation on Degenerative Discus Disease Patients (Clinical Trial)
Brief Title: Effectiveness and Safety of Mesenchymal Stem Cell (MSC) Implantation on Degenerative Discus Disease Patients
Acronym: MSC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmad Jabir Rahyussalim (Other)
Responsible Party: Sponsor-Investigator, Ahmad Jabir Rahyussalim, Dr. dr. Rahyussalim SpOT(K), Indonesia University
Organization: Indonesia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-02-0143
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Degenerative Disc Disease; Low Back Pain; Disc Degeneration
Keywords: DDD; MSC
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stem Cell (Experimental): Mesenchymal Stem cell + Nacl 0.9%
  Interventions: Drug: Mesenchymal Stem Cell + NaCl 0,9% 2ml

INTERVENTIONS:
Drug: Mesenchymal Stem Cell + NaCl 0,9% 2ml — Patients enrolled in Cipto Mangunkusumo Hospital with degenerative disc disease with no promising result after conventional treatment.

SUMMARY:
This study evaluates the effectivity and safety of MSC implantation on Degenerative Disc Disease Patients by assessing visual analog scale, ROM improvement and MRI examination.

DETAILED DESCRIPTION:
The team plan to conduct research to look at the effectiveness and safety of mesenchymal stem cell implantation therapy in intervertebral disc degeneration patients.

The use of allogenic mesenchymal stem cells from the umbilical cord was chosen because patients with degeneration of the intervertebral disc are elderly (over 50 years old) so that autologous mesenchymal stem cell administration is not possible in terms of taking the source of cells (bone marrow) nor the quality of mesenchymal stem cells obtained.

This study will assess the improvement of clinical symptoms (VAS to assess pain scale, ASIA and Frankel scale, as well as assessment of the widening of the lumbar region using the Schober Test), changes in the structure of the intervertebral discs (through MRI examination and grading the degree of intervertebral disc degeneration), conduction function spinal cord nerve (somatosensory evoked potential / SSEP), myelography / EMG, and assessment of the quality of life status of patients using the Oswestry Disability Index.

ELIGIBILITY:
Inclusion Criteria:

1. Patients enrolled in Cipto Mangunkusumo Hospital with degenerative disc disease with no promising result after conventional treatment.
2. No history of metabolic, autoimun and genetic disease(s).
3. No active infection (HbsAg, HIV, CMV, Rubella).
4. Agree to participate the study by signing informed consent form.

Exclusion Criteria:

1. Patients under 20 years old.
2. Declined to participate in the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-07-24 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of Low Back Pain | 6 months
  Evaluates pain quality using Visual Analog Scale (VAS) from 0 - 10. Zero is no pain at all, one is the the least pain and ten is the most painful. The numbers are expected to be lower after MSC implantation.
Tissue Improvement | 6 months
  Tissue improvement confirmed by intervertebral disc MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia